CLINICAL TRIAL: NCT00004896
Title: Phase II Study of High-Dose Busulfan and Cyclophosphamide Followed by Allogeneic Bone Marrow Transplantation for Patients With Acute Myelogenous Leukemia
Brief Title: Busulfan and Cyclophosphamide Followed by Bone Marrow Transplantation in Treating Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: NU 91H4T; NU-91H4T; NCI-G00-1686
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; adult acute monocytic leukemia (M5b); previously treated myelodysplastic syndromes; myelodysplastic/myeloproliferative disease, unclassifiable; atypical chronic myeloid leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Congenital Abnormalities | interventions — Busulfan; Cyclophosphamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Procedure: allogeneic bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with donor bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of busulfan and cyclophosphamide followed by bone marrow transplantation in treating patients who have acute myelogenous leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the remission duration, disease-free survival, and overall survival of patients with acute myelogenous leukemia in remission or early relapse or myelodysplastic syndrome treated with high-dose busulfan and cyclophosphamide followed by allogeneic bone marrow transplantation.

OUTLINE: Patients receive oral high-dose busulfan every 6 hours for 14-16 doses on days -9 to -6, followed by high-dose cyclophosphamide IV over 1 hour on days -5 to -2. Allogeneic bone marrow is infused on day 0.

Patients who have already had 1 transplant receive high-dose cyclophosphamide IV on days -6 and -5, total body irradiation twice a day on days -4 to -1, and allogeneic bone marrow infusion on day 0.

All patients receive prophylaxis for graft versus host disease.

Patients are followed every 6 months for at least 2 years.

PROJECTED ACCRUAL: A total of 25-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically proven (from bone marrow aspirate smears or touch preps of marrow biopsy) acute myelogenous leukemia or myelodysplastic syndrome of 1 of the following subtypes:

  * Acute myeloblastic leukemia (M1, M2)
  * Acute promyelocytic leukemia (M3)
  * Acute myelomonocytic leukemia (M4)
  * Acute monocytic leukemia (M5)
  * Acute erythroleukemia (M6)
  * Acute megakaryocytic leukemia (M7)
  * Refractory anemia
  * Refractory anemia with excess blasts
  * Refractory anemia with excess blasts in transformation
  * Refractory anemia with ringed sideroblasts
  * Chronic myelomonocytic leukemia
* In remission or in early relapse as defined by less than 20% blast cells in the marrow or overt active acute myeloid leukemia
* Suitable marrow donor, defined as a sibling donor matched at the HLA-A, HLA-B, and HLA-D/DR locus nonreactive in bidirectional mixed lymphocyte culture or a donor who is mismatched at 1 antigen loci
* Active CNS disease allowed

PATIENT CHARACTERISTICS:

Age:

* 16 to physiologic 60

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN) unless due to Gilbert's disease
* SGOT no greater than 3 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* Cardiac ejection fraction normal

Pulmonary:

* FEV_1 at least 50% of predicted
* DLCO at least 50% of predicted

Other:

* HIV negative
* No evidence of persistent infection
* No concurrent organ damage or medical problems that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent antibiotics

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-10; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Tallman, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States